CLINICAL TRIAL: NCT04952129
Title: Randomised Phase Ib Trial to Determine the Optimal Selenium Status to Prevent Colorectal Adenoma Recurrence: OSCAR
Brief Title: Optimal Selenium for Bowel Polyps (OSCAR)
Acronym: OSCAR
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Auckland, New Zealand (Other)
Collaborators: Cancer Trials New Zealand (Other); Counties Manukau Health (Other); Waikato Hospital (Other)
Responsible Party: Principal Investigator, Michael Jameson, Associate Professor, University of Auckland, New Zealand
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: OSCAR
Record Dates: First submitted 2021-06-14; First posted 2021-07-07 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Colorectal Adenoma
Keywords: selenium; colorectal adenoma; selenomethionine; methylselenocysteine; selenoprotein P
MeSH Terms: interventions — Selenomethionine; Selenium; selenomethylselenocysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Selenomethionine (Experimental): 50 micrograms of selenium as Selenomethionine per oral capsule. Dosage: One capsule a day for 6 weeks, followed by two capsules per day for 6 weeks.
  Interventions: Drug: Selenomethionine
- Methylselenocysteine (Experimental): 50 micrograms of selenium as Methylselenocysteine per oral capsule. Dosage: One capsule a day for 6 weeks, followed by two capsules per day for 6 weeks.
  Interventions: Drug: Methylselenocysteine

INTERVENTIONS:
Drug: Selenomethionine — Seleno-amino acid
  Other Names: L-selenomethionine
  Arms: Selenomethionine
Drug: Methylselenocysteine — Seleno-amino acid
  Other Names: Se-methyl-selenocysteine
  Arms: Methylselenocysteine

SUMMARY:
New Zealand (NZ) has high bowel cancer rates, which the Bowel Screening Programme aims to reduce by early detection of bowel cancer and its precursor, adenomas (polyps). Bowel cancer and adenoma rates are higher in countries like NZ with low intake of the essential trace mineral selenium. Overseas, trials of selenium supplements reduced adenoma recurrence in people with low blood selenium, but not with high levels (where adding selenium increased health risks). Laboratory research explained this, and found certain types of selenium are safer and more effective. The optimal type and dose of selenium to use in NZ cancer prevention trials is not known.

The goal of this clinical trial is to find out how to achieve the optimal amount of body selenium in people who have had a high risk bowel adenoma removed. The main questions it aims to answer are:

* what dose of selenium taken by mouth will maximise levels of the main selenium protein in blood;
* whether one type of organic selenium is better than the other at increasing blood levels of this selenium protein;
* whether a larger dose of selenium is needed in people who start with lower blood selenium levels;

Participants will take one selenium capsule a day for 6 weeks then two capsules a day for 6 weeks. Each participant will have blood tests at baseline, then blood tests and evaluation of side effects at 6 weeks and 12 weeks.

Researchers will compare these results in the participants taking each type of selenium (selenomethionine or methylselenocysteine).

DETAILED DESCRIPTION:
The main aim of this trial is to evaluate which dose and type of selenium (Se), either selenomethionine or methylselenocysteine, achieves optimal selenium status, in order to maximise its potential for cancer prevention without causing health problems from excessive Se intake. The trial will also evaluate how much Se is needed according to Se blood levels before starting Se in the trial, adverse events and recruitment rates.

This trial will recruit 60 participants from Middlemore and Waikato Hospitals with at least one advanced colorectal adenoma removed through the Bowel Screening Programme. Participants will be randomised (1:1) to take either selenomethionine or methylselenocysteine, dosed at Se 50 mcg/day for 6 weeks then 100 mcg/day for 6 weeks.

Co-primary objectives:

To determine whether:

1. Se 50 µg/day for 6 weeks significantly increases plasma selenoprotein P (SEPP) from baseline;
2. the increase in plasma SEPP from baseline is greater with Se 100 µg/day than 50 µg/day only when baseline plasma Se is below the median value for the trial population;
3. the increase in plasma SEPP from baseline is not different between MSC and SLM at each dose level.

Secondary objectives:

To determine:

1. change in plasma Se levels by Se type and dose;
2. change in white blood cell DNA damage from baseline by Se type and dose;
3. feasibility (assessed by recruitment rates, adverse events, compliance with trial medication and participant experience).

Trial assessments:

* blood tests at baseline, then 6 weeks and 12 weeks after initiating Se dosing;
* adverse events and trial medication compliance assessed 6 weeks and 12 weeks after initiating Se dosing;
* participant experience survey on completion of trial medication dosing.

ELIGIBILITY:
Inclusion Criteria:

Participants will have all of the following:

* pathologically-confirmed advanced adenoma (defined as any one of >/= 10mm diameter, >/= 3 adenomas, high-grade dysplasia, tubulovillous or villous adenoma) 5 diagnosed at first colonoscopy in the National bowel screening programme within the previous 6 months;
* no residual colorectal adenomas;
* next colonoscopy planned within 5 years;
* willing and able to comply with all trial requirements, including treatment and assessments;
* signed written, informed consent.

Exclusion Criteria:

Participants will have none of the following:

* currently taking selenium supplements (including in multivitamins) or within the last 6 weeks;
* previous history of colorectal adenoma, colorectal cancer or familial colorectal cancer syndrome;
* other significant cancers within the last 5 years;
* concurrent medical conditions that, in the opinion of the investigators, would compromise either participant safety or the integrity of the data (e.g., malabsorption);
* male participants with a female partner of childbearing potential or pregnant, and unwilling to remain abstinent or use effective contraception (including barrier contraception with a pregnant partner).

Ages: 60 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2022-05-06 (Actual); Primary Completion 2023-12-11 (Actual); Study Completion 2023-12-11 (Actual)

PRIMARY OUTCOMES:
Plasma SEPP1 concentration 1 | At 6 weeks
  To determine whether 50 micrograms/day of selenium for 6 weeks significantly increases plasma SEPP1 from baseline.
Plasma SEPP1 concentration 2 | At 6 and 12 weeks
  To determine whether the change in plasma SEPP1 from baseline is greater with selenium 100 micrograms/day than 50 micrograms/day only when baseline plasma selenium is below the median value for the trial population.
Plasma SEPP1 concentration 3 | At 6 and 12 weeks
  To determine whether the change in plasma SEPP1 from baseline is not different between methylselenocysteine and selenomethionine at each dose.

SECONDARY OUTCOMES:
Plasma selenium | At 6 and 12 weeks
  To determine change in plasma selenium levels by selenium type and dose.
Treatment-emergent adverse effects | At all time points
  To determine the incidence of treatment-emergent adverse effects as classified according to NCI-CTCAE version 5.0
White blood cell DNA damage | At 6 and 12 weeks
  To determine change in DNA damage (relative to baseline) by selenium type and dose.
Recruitment | At baseline
  To determine to percentage of subjects who after being offered the study continue on to study entry.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Jameson, PhD, Principal Investigator — University of Auckland, New Zealand
Locations (2):
- New Zealand (2):
  - Waikato DHB, Hamilton, Waikato Region
  - Counties Manukau DHB, Auckland

IPD SHARING:
Plan to Share IPD: No